CLINICAL TRIAL: NCT00458861
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy, Safety, PK, and PD of BG9924 When Given in Combo With MTX to Subjects With Active RA Who Have Had an Inadequate Response to Anti-TNF
Brief Title: BG9924 in Combination With Methotrexate for Participants With Active Rheumatoid Arthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis of data failed to meet primary endpoint.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 104RA203; 2006-005467-26 (EudraCT Number)
Record Dates: First submitted 2007-03-22; First posted 2007-04-11 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2015-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Active Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BG9924 (Experimental): Subcutaneous administration of BG9924 given every other week for 12 weeks
  Interventions: Biological: BG9924
- Placebo (Placebo Comparator): Subcutaneous administration of placebo given every other week for 12 weeks
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Biological: BG9924 — Subcutaneous administration of BG9924 given every other week for 12 weeks
  Arms: BG9924
Other: Placebo Comparator — Subcutaneous administration of placebo given every other week for 12 weeks
  Arms: Placebo

SUMMARY:
This Phase 2b study is designed to evaluate the efficacy and safety of BG9924 given subcutaneously (SC) versus placebo in participants with active rheumatoid arthritis (RA) who have previously had an inadequate response to treatment with anti-tumor necrosis factor (anti-TNF) therapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of rheumatoid arthritis (functional class I - III) at least 6 months prior to baseline
* Methotrexate (10 mg/week to 25 mg/week) > 3 months prior to Day 0 (stable dose > 4 weeks prior to Day 0)
* Must have had an inadequate response to anti-TNF therapy due to inadequate efficacy

Key Exclusion Criteria:

Medical History

* Serious local infection or systemic infection within 3 months of Day 0
* History (Hx) of recurrent infections requiring oral or parental anti-infective treatment
* Hx of tuberculosis (TB) or positive purified protein derivative (PPD) test during the screening period

Laboratory Tests

* Clinically significant lab tests at screening; or
* Positive for hepatitis C antibody or hepatitis B at screening

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2007-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Evaluate efficacy of BG9924 in combination with methotrexate in RA participants who have had an inadequate response to anti-TNF therapy | 26 weeks

SECONDARY OUTCOMES:
Assess the safety and tolerability of BG9924 in this participant population. | 26 weeks
Assess the pharmacokinetic and pharmacodynamic profile of BG9924 in this participant population. | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Stanford University, Palo Alto, California, United States